CLINICAL TRIAL: NCT02089490
Title: Prospective Follow-up Study for the Evaluation of the Safety and Efficacy of the Dermal Substitute NEVELIA® in the Treatment of Third-degree Burns and Reconstructive Surgery
Brief Title: Evaluation of NEVELIA® in Terms of Safety and Efficacy for Third-degree Burns Treatment or Reconstructive Surgery
Acronym: NEVAL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Symatese (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCS2 NEVELIA
Record Dates: First submitted 2014-03-14; First posted 2014-03-17 (Estimated); Last update posted 2014-03-17 (Estimated); Status verified 2014-03

CONDITIONS: Third-degree Burns; Reconstructive Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- NEVELIA® (Experimental): NEVELIA® implantation according to the intended use in the leaflet, prior to autologous skin grafting planned 3 weeks after its application.
  Interventions: Device: NEVELIA® implantation

INTERVENTIONS:
Device: NEVELIA® implantation — Skin substitute implantation followed by ultra-thin epidermal graft
  Other Names: Skin substitute graft; Skin substitute placement

SUMMARY:
The dermal substitute NEVELIA® has received CE marking in July 9, 2013. Its use in the NEVAL protocol will be in accordance with its leaflet, i.e. for the treatment of burns or in case of reconstructive plastic surgery.

The matric implantation will be followed by autologous skin grafting when the neodermis formation will be observed.

DETAILED DESCRIPTION:
The NEVAL protocol is a descriptive study conducted in order to confirm the clinical evidence of safety and performance of NEVELIA®, as described in the literature on equivalent products.

This dermal substitute consists of an inner biodegradable dermal substitute made of bovine collagen (collagen of type I), covered with an outer silicone membrane. Its porosity and the speed of degradation allow the act of recolonization by the fibroblasts and initiation of the vascularization process within 3 weeks. The application procedure requires removement of the silicone layer and wound covering with an ultra-thin epidermal graft, possibly meshed. This surgical procedure is well-known and permits an ultra-thin epidermal graft.

All the patients will be treated with NEVELIA®, prior to autologous skin grafting within 3 weeks after its application. Then, three follow-up visits will be planned: post operatively, at 6 and 12 months.

The objectives are:

* Primary objective: To assess the type and frequency of complications
* Secondary objectives:

  * To assess the take rate of NEVELIA®
  * To assess the take rate of skin graft
  * To assess the satisfaction rate of physician and patient,
  * To assess the quality of the healed skin,
  * To assess the rate of re-operation at 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 or older
* Patient geographically stable,
* Patient requiring dermal reconstruction after third-degree burns, reconstructive surgery or trauma surgery;
* Patient who signed the non-opposition form;
* Patient able to be followed up to 12 months.

Exclusion Criteria:

* Patient with clinical signs of wound infection;
* Allergic patient or with known allergy to bovine collagen or silicone;
* Patient with life-threatening conditions;
* Patient receiving a treatment that may affect wound healing;
* Patient with an autoimmune or immunosuppressive disease;
* Patient with a suspected neurological disease as Creutzfeldt-Jakob disease;
* Patient simultaneously participating in another study;
* Pregnant or nursing woman.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2014-04; Primary Completion 2016-01 (Estimated); Study Completion 2016-04 (Estimated)

PRIMARY OUTCOMES:
Assessment of the type and frequency of complications related to NEVELIA® | Up to 12 months

SECONDARY OUTCOMES:
Take rate of NEVELIA® | At Day 21
Take rate of skin graft | At Day 28, 6 and 12 months
Satisfaction rate of physician and patient | At 6 and 12 months
Quality of healed skin | At 6 and 12 months
  Vancouver score
Re-operation rate | At 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Casoli, MD PhD, Principal Investigator — Centre François Xavier Michelet - CHU de Bordeaux, FRANCE
Locations (1):
- Centre François Xavier Michelet - CHU de Bordeaux, Bordeaux, France

REFERENCES:
- [Background] Shevchenko RV, James SL, James SE. A review of tissue-engineered skin bioconstructs available for skin reconstruction. J R Soc Interface. 2010 Feb 6;7(43):229-58. doi: 10.1098/rsif.2009.0403. Epub 2009 Oct 28. PMID 19864266
- [Background] Clark RA, Ghosh K, Tonnesen MG. Tissue engineering for cutaneous wounds. J Invest Dermatol. 2007 May;127(5):1018-29. doi: 10.1038/sj.jid.5700715. PMID 17435787
- [Background] MacNeil S. Progress and opportunities for tissue-engineered skin. Nature. 2007 Feb 22;445(7130):874-80. doi: 10.1038/nature05664. PMID 17314974
- [Background] Pham C, Greenwood J, Cleland H, Woodruff P, Maddern G. Bioengineered skin substitutes for the management of burns: a systematic review. Burns. 2007 Dec;33(8):946-57. doi: 10.1016/j.burns.2007.03.020. Epub 2007 Sep 7. PMID 17825993
- [Background] Koenen W, Felcht M, Goerdt S, Faulhaber J. Skin substitutes in dermatosurgery. G Ital Dermatol Venereol. 2010 Oct;145(5):637-49. PMID 20930698
- [Background] Chaouat M, Zakine G, Mimoun M. [Principles of the local treatment: Surgical processing]. Pathol Biol (Paris). 2011 Jun;59(3):e57-61. doi: 10.1016/j.patbio.2009.12.003. Epub 2010 Feb 8. French. PMID 20116939